CLINICAL TRIAL: NCT06374303
Title: Novel Intervention to Improve Food Insecurity Among Individuals With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Professor, PI, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS 00001940
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Food Security
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-groups pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Education (NE) control condition (No Intervention): Nutritional Education (NE) participants received brief education, a list of FI-related resources in their community, and assistance with contacting those resources.
- Nutritional Eduction + Meal Delivery (NE+MD) experimental condition (Experimental): NE + Meal Delivery (NE+MD) participants received the same educational platform plus weekly meal deliveries using a commercial service that delivers premade, refrigerated meals directly to the participant's home.
  Interventions: Other: NE + Meal Delivery (NE+MD) intervention

INTERVENTIONS:
Other: NE + Meal Delivery (NE+MD) intervention — NE + Meal Delivery (NE+MD) participants received the same educational platform plus weekly meal deliveries using a commercial service that delivers premade, refrigerated meals directly to the participant's home.
  Arms: Nutritional Eduction + Meal Delivery (NE+MD) experimental condition

SUMMARY:
The adverse consequences of illicit opioid use (e.g., overdose, premature death) are the focus of intensive research efforts. However, other serious health problems among individuals with opioid use disorder (OUD) have received far less attention. Food insecurity (FI) is 4-7 times greater among individuals with OUD than the general population. In addition to the increased healthcare utilization and costs, poor health outcomes, and adverse social consequences associated with FI in the general population, patients with co-occurring FI and OUD are at increased risk for licit and illicit drug use, sexual and drug risk behaviors, infectious disease, and a two-fold greater odds of premature death.

In this randomized pilot study, we evaluated a novel, mail-based meal delivery intervention for improving household FI and other outcomes among individuals receiving methadone or buprenorphine maintenance for OUD.

Fifty adults with FI and OUD were randomized to one of two 12-week experimental conditions: Nutritional Education (NE) participants received brief education, a list of FI-related resources in their community, and assistance with contacting those resources. NE + Meal Delivery (NE+MD) participants received the same educational platform plus weekly meal deliveries using a commercial service that delivers premade, refrigerated meals directly to the participant's home.

The primary outcome of household FI was measured at monthly assessments using the USDA Household Food Security Survey. Secondary measures included depression symptoms (Beck Depression Inventory), quality of life (RAND-36 Quality of Life Survey), and drug use as measured by biochemical urinalysis.

The NE+MD intervention was associated with significant improvements in household FI, with fewer NE+MD participants meeting criteria for FI vs. NE participants at all three assessment timepoints (p's<.05). Retention rates were similar between the two groups (88% and 84% for NE+MD and NE conditions, respectively; p=.68). Intervention acceptability was also high, with NE+MD participants rating the enjoyment and convenience of the meals at 81 and 93, respectively (range: 0-100).

Changes in FI status were also associated with improvements in other areas of functioning. NE+MD participants experienced reductions in depression symptomatology, with Beck Depression Inventory scores lower than intake at Weeks 4 and 8 (p's<.05) and no changes among NE participants. NE+MD participants also experienced improvements on four of the eight subscales of the RAND-36 Quality of Life Health Survey (i.e., General Health, Bodily Pain, Mental Health, Role Emotional; p's<.05), with no changes among NE participants.

This study represents the first effort to develop and evaluate a novel intervention to reduce FI and related problems among individuals with OUD. These pilot data support the feasibility, acceptability and initial efficacy of the NE+MD intervention for improving household FI, as well as provide exciting new preliminary evidence suggesting that FI may be linked to participants' mental and physical health.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* receiving methadone or buprenorphine treatment for OUD
* meet criteria for current FI as measured by the 18-item US Household Food Security Survey (FSS; Economic Research Service, USDA, 2012)

Exclusion Criteria:

* Significant psychiatric or medical illness
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Household food insecurity Survey | 3 month study duration
  measured using the USDA Household Food Security

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Sigmon, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No